CLINICAL TRIAL: NCT01070875
Title: Partial Thromboplastin Time During the First 24 Hours of Antithrombotic Prophylaxis Using Unfractionated Heparin: Comparison of a 2 Times Per Day Versus Per 3 Times a Day Dosage
Brief Title: Partial Thromboplastin Time During the First 24 Hours of Antithrombotic Prophylaxis Using Unfractionated Heparin (UFH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NM 2010-002
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Thrombosis
Keywords: Antithrombotic prophylaxis
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- UFH 5000 U three times per day (Active Comparator): Study subjects will be randomized to receive unfractionated heparin 5000 U subcutaneous three times a day.
  Interventions: Drug: Variation of heparin dose
- UFH 5000 U two times per day (Active Comparator): Study subjects will be randomized to receive unfractionated heparin 5000 U subcutaneous two times a day.
  Interventions: Drug: Variation of heparin dose

INTERVENTIONS:
Drug: Variation of heparin dose — Study subjects will be randomized to receive unfractionated heparin 5000 U subcutaneous two times a day.
  Arms: UFH 5000 U two times per day
Drug: Variation of heparin dose — Study subjects will be randomized to receive heparin 5000 U subcutaneous three times a day.
  Arms: UFH 5000 U three times per day

SUMMARY:
This study is designed to assess the incidence of abnormal partial thromboplastin time in patients receiving unfractionated heparin (UFH) 5000 U 2 times a day versus 3 times a day.

The basic hypothesis of this study is that patients receiving UFH 5000 U subcutaneously 3 times a day will have a higher proportion of elevated partial thromboplastin time than patients receiving UFH 5000 U subcutaneously twice a day.

DETAILED DESCRIPTION:
Administration of subcutaneous UFH for antithrombotic prophylaxis is standard therapy in the postoperative setting. Often, a dosage of 5000 U twice a day has been used, with a demonstrated antithrombotic efficacy and an acceptable hemorrhagic complication profile. However, recent surgery guidelines regarding antithrombotic prophylaxis with UFH 5000 U suggest that a thrice daily regimen should be used following major oncologic surgeries. These new guidelines have raised some concerns in anaesthesiology, particularly regarding the safety of epidural catheters combined with thrice daily heparin. Optimal analgesia during the early postoperative period following some types of major oncologic surgery involves the placement of epidural catheters. Epidural analgesia provides the best relief of the significant pain which may be present after thoracotomy or supraumbilical laparotomy during the early postoperative period, improving ambulation, coughing, pulmonary function, bowel function as well as short and long-term quality of life. However, the benefits of epidural catheters must outweigh the risk of complications, the most feared being spinal hematoma. Recent guidelines in anaesthesiology support the placement of epidural catheters with the concomitant administration of UFH 5000 U two times a day. However, these guidelines do not clearly support the placement of an epidural catheter if a three times a day regimen is used, very little data being available to assess the risk of this practice. Older studies (1973) suggest that a significant proportion of patients (15%) will develop abnormal partial thromboplastin times using a three times a day regimen. However, it is not known if these results are still consistent with more recent laboratory technologies, or how they compare to twice daily heparin. In the absence of even basic data regarding systemic effect on coagulation, it is difficult at this time to begin to determine safe practice regarding the placement of an epidural catheter in presence of a three times a day UFH 5000 U regimen. This study is designed to obtain this data.

Methods: As needed for standard anesthesia , surgical and post-operative care, an arterial line will be placed and kept for the first 24 hours postoperatively. Immediately prior the first UFH dose and hourly for the following 24 hours, blood samples for partial thromboplastin times will collected through the arterial line. The first dose of UFH will be given in the operating room by the anaesthesiologist. A blood sample for partial thromboplastin time will also be collected 3 days following the first dose of UFH.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or older
* Patients undergoing an elective thoracic surgery requiring the placement of an arterial line and antithrombotic prophylaxis

Exclusion Criteria:

* Pre-existing coagulopathy
* Severe renal failure
* Known allergy to heparin
* History of heparin induced thrombocytopenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2010-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
To determine the proportion of abnormal partial thromboplastin time values during the first 24 hours of antithrombotic prophylaxis in patients receiving UFH 5000 U 2 times a day versus 3 times a day following surgery. | 24 hours starting at time of first dose of heparin

SECONDARY OUTCOMES:
To describe the changes over time of the partial thromboplastin time during the first 24 hours following the administration of UFH. | 24 hours starting at time of first dose of heparin
To assess a possible relationship between coagulation abnormalities and demographic, biological or physical variables. | 24 hours starting at time of first dose of heparin
To determine the proportion of abnormal partial thromboplastin time values 3 days after the administration of the first dose of UFH 5000 U 2 times versus 3 times a day. | Three days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Massicotte, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal-Hôpital Notre-Dame, Montreal, Quebec, Canada